CLINICAL TRIAL: NCT06021197
Title: NMDA-enhancing Treatment for Cognitive Dysfunction of Schizophrenia Patients During Symptomatic Remission
Brief Title: NMDA-enhancing Treatment for Cognitive Dysfunction of Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMUH111-REC3-228
Record Dates: First submitted 2023-08-28; First posted 2023-09-01 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NMDA; Symptomatic remission
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMDAE (Experimental): An NMDA enhancer
  Interventions: Drug: NMDAE
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Cap

INTERVENTIONS:
Drug: NMDAE — Use of an NMDA enhancer for the treatment of CIAS
  Arms: NMDAE
Drug: Placebo Cap — Use of placebo as a comparator
  Arms: Placebo

SUMMARY:
Cognitive impairment, the core psychopathology of schizophrenia, usually persists in schizophrenia patients even during symptomatic remission. While cognitive impairment associated with schizophrenia (CIAS) is an important therapeutic target, hypofunction of N-methyl-D-aspartate receptor (NMDAR) is a key factor of CIAS. This study aims to examine the efficacy and safety of an NMDA-enhancer (NMDAE) for the treatment of CIAS in schizophrenia patients during symptomatic remission.

DETAILED DESCRIPTION:
Cognitive impairment, the core psychopathology and the outcome determinant of schizophrenia, usually persists in schizophrenia patients even during symptomatic remission. Cognitive impairment associated with schizophrenia (CIAS) is an important therapeutic target; and hypofunction of N-methyl-D-aspartate receptor (NMDAR) is a key factor of CIAS. Whether NMDAR-enhancing treatment can truly improve cognitive function needs to be tested in schizophrenia patients during symptomatic remission. This study aims to examine the efficacy and safety of an NMDA-enhancer (NMDAE) for the treatment of CIAS in schizophrenia patients during symptomatic remission.

The subjects are the patients with schizophrenia during symptomatic remission. They keep their original treatment and are randomly, double-blindly assigned into two treatment groups for 12 weeks: (1) NMDAE, or (2) placebo. At weeks 0 and 12, 7 cognitive domains will be measured. At weeks 0, 4, 8, and 12, Global Assessment of Function, Quality of Life Scale, various clinical-symptom rating scales, and side effects scales will be measured too.

Chi-square (or Fisher's exact test) will be used to compare differences of categorical variables and t-test (or Mann-Whitney test if the distribution is not normal) for continuous variables between treatment groups. Mean changes from baseline in repeated-measure assessments will be assessed using the generalized estimating equation (GEE). All p values for clinical measures will be based on two-tailed tests with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Have a Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, Text Revision (DSM-5 -TR) diagnosis of schizophrenia
* Fulfill the Remission in Schizophrenia Working Group (RSWG) criteria for remission (Andreasen et al., 2005): each of eight items (delusions, unusual thought content, hallucinatory behavior, conceptual disorganization, mannerisms/posturing, blunted affect, passive/apathetic social withdrawal, and lack of spontaneity and flow of conversation) in the Positive and Negative Syndrome Scale (PANSS) (Kay et al., 1987) scoring 3 or lower for 6 months or longer; in addition, have a baseline total score of 59 or lower in the PANSS
* Are physically healthy and laboratory assessments (including blood routine, biochemical tests) are clinically insignificant;
* Have been keeping a fixed dose of antipsychotics (excluding clozapine) for at least 6 months, and that is not allowed to change during the 12-week study period
* Have sufficient education to communicate effectively and are capable of completing the assessments of the study
* Agree to participate in the study and provide written informed consent

Exclusion Criteria:

* DSM-5-TR diagnosis of intellectual disability or substance (including alcohol) use disorder
* History of epilepsy, head trauma, or serious medical or central nervous system diseases (other than schizophrenia) which may interfere with the study
* Pregnancy or lactation
* Inability to follow protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change of cognitive function composite | Week 0, 12
  Ten tests for assessment of 7 cognitive domains:
  1. speed of processing (assessed by Category Fluency, Trail Marking A, Wechsler Adult Intelligence Scale(WAIS)-III Digit Symbol-Coding)
  2. sustained attention (Continuous Performance Test)
  3. working memory: verbal (digit span) and nonverbal (spatial span)
  4. verbal learning and memory (WMS-III, word listing)
  5. visual learning and memory (WMS-III, visual reproduction)
  6. reasoning and problem solving (WISC-III, Maze)
  7. social cognition (MSCEIT Version 2)
  For the domain (a. and c.) with more than one test, a composite T score will be calculated by standardizing the average of each T score. Furthermore, a global composite score (for all seven domains) and a neurocognitive composite score (for the first 6 domains) will be also calculated by standardizing the average of the T score (Lane HY et al, JAMA Psychiatry 2013)

SECONDARY OUTCOMES:
Change of Global Assessment of Functioning composite | week 0, 4, 8, 12
  Assessment of social, occupational, and psychological function. Minimum value: 1, maximum value:100, the higher scores mean better function.
Change of Quality of Life Scale | week 0, 4, 8, 12
  Assessment of life quality. Minimum value: 0, maximum value:126, the higher scores mean a better outcome.

OTHER OUTCOMES:
Change of Positive and Negative Syndrome Scale (PANSS) | week 0, 4, 8, 12
  Assessment of overall symptoms. Minimum value: 30, maximum value:210, the higher scores mean a worse outcome.
Change of scales for the Assessment of Negative Symptoms (SANS) total score | week 0, 4, 8, 12
  Assessment of negative symptoms. Minimum value: 0, maximum value:100, the higher scores mean a worse outcome.
Change of Positive subscale of PANSS | week 0, 4, 8, 12
  Assessment of positive symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
Change of Negative subscale of PANSS | week 0, 4, 8, 12
  Assessment of negative symptoms. Minimum value: 7, maximum value:49, the higher scores mean a worse outcome.
Change of General Psychopathology subscale of PANSS | week 0, 4, 8, 12
  Assessment of general psychopathology. Minimum value: 16, maximum value:112, the higher scores mean a worse outcome.
Change of Clinical Global Impression | week 0, 4, 8, 12
  Assessment of general impression. Minimum value: 1, maximum value:7, the higher scores mean a worse outcome.
Change of Hamilton Rating Scale for Depression | week 0, 4, 8, 12
  Assessment of depressive symptoms. Minimum value: 0, maximum value:52, the higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, China Medical University Hospital, Taichung, Taiwan